CLINICAL TRIAL: NCT02468011
Title: Whole Body Vibration Induced Muscle Activity in Different Position of Lower Extremity: Effect of the Changes in Length of Soleus Muscle and Angle of Ankle
Brief Title: Whole Body Vibration Induced Muscle Activity and Effect of the Changes in Length of Soleus Muscle and Angle of Ankle
Acronym: WBVIMR-SL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ilhan Karacan, Clinical Associated Professor, Head of department, Bagcilar Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BEAH FTR-10
Record Dates: First submitted 2015-06-08; First posted 2015-06-10 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Muscle Physiology
MeSH Terms: interventions — Vibration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vibration (Experimental): Whole body vibration with 35 Hz
  Interventions: Other: vibration

INTERVENTIONS:
Other: vibration — vibration will be applied at 35 Hz

SUMMARY:
Previous studies reported that myoelectrical activity increased during whole body vibration (WBV). The investigators hypothesized that the change in soleus muscle length does not affect the whole body vibration induced soleus reflex muscle activity but the change in ankle angle affects the whole body induced soleus reflex muscle activity. The purpose of this study is to test this hypothesis.

DETAILED DESCRIPTION:
Eighteen healthy young adult men are planned to include in this study. Surface electrodes will be placed on the right soleus muscle's belly. The electrodes (10-mm in diameter, inter-electrode distance of 20 mm) were arranged in the direction of the muscle fibers. The skin overlying the muscle was shaved, light abrasion was applied, and the skin was cleaned using 70% alcohol.

A piezo-electric accelerometer (LIS344ALH full-scale of ±6 g linear accelerometer, ECOPACK) will be placed on the achilles tendon and a force sensor (FC2331-0000-2000L Compression Load Sensor, France) will be placed under the right heel. All data will be recorded by PowerLab (data acquisition system, ADInstruments, Australia) device. The data were processed offline with a computer. All surface electromyography (SEMG) analyses were conducted using a software (LABCHART7 ver. 7.3.3; POWERLAB System, ADInstruments). All SEMG recordings were 80-500 Hz band-pass filtered. Root-mean-square values (RMS) were calculated from the filtered SEMG signal.

WBV (PowerPlate Pro5) with high amplitude at 35 Hz will be applied. Participants were barefooted, and no sponge or foam was placed between the vibration platform and their feet. Participants will stand in different position with their knees locked during WBV. Their hips and knees were in a neutral position. Positions: Position-1: Upright standing on zero sloping vibration platform Position-2: Standing with 10 degrees ankle dorsiflexion on zero sloping vibration platform Position-3: Standing with 20 degrees ankle plantarflexion on zero sloping vibration platform Position-4: Upright standing on twenty degrees forward inclined vibration platform (angle angle will be 20 degrees ankle plantarflexion) Position-5: Leaning forward while standing on twenty degrees forward inclined vibration platform (angle angle will be neutral) Position-6: Upright standing on 10 degrees backward inclined vibration platform (angle angle will be 20 degrees ankle dorsiflexion) Position-7: Leaning backward while standing on 10 degrees backward inclined vibration platform (angle angle will be neutral) Sequence of the position will be random. Maximal voluntary contraction (MVC) was determined for each subject at the beginning of each position using magnitude of force between heel and vibration platform the when the subject attempted to activate the soleus muscle maximally. Then vibration exposure will be 30 seconds.

The participants were instructed to relax their muscles throughout the recordings during WBV and were trained using electromyographic feedback to this end. WBV may impair the sense of balance and muscles may be activated to restore balance. To overcome this problem, the participants were familiarized with WBV with a 15 s trial session on the WBV device and they were asked to use the handles of the device to secure their balance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men
* Men with ages varying between 20 and 40 years
* Right-handed men

Exclusion Criteria:

* Bone, muscle/tendon, joint, vascular, dermatologic diseases in lower extremities and spine
* Medication that could affect the musculoskeletal system
* Postural abnormalities (scoliosis, kyphosis, etc)
* Systemic diseases (Cardiopulmonary diseases, diabetes mellitus etc)
* Obesity (BMI>30 kg/m2)
* Vertigo / dizziness

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-06; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Vibration induced reflex muscle activity level | Four months

CONTACTS AND LOCATIONS:
Overall Officials: 90 212 4404000 90 212 4404000, MD, Study Chair — Bagcilar Training & Research Hospital

REFERENCES:
- [Background] Pollock RD, Woledge RC, Martin FC, Newham DJ. Effects of whole body vibration on motor unit recruitment and threshold. J Appl Physiol (1985). 2012 Feb;112(3):388-95. doi: 10.1152/japplphysiol.01223.2010. Epub 2011 Nov 17. PMID 22096119
- [Background] Ritzmann R, Kramer A, Gollhofer A, Taube W. The effect of whole body vibration on the H-reflex, the stretch reflex, and the short-latency response during hopping. Scand J Med Sci Sports. 2013 Jun;23(3):331-9. doi: 10.1111/j.1600-0838.2011.01388.x. PMID 23802287
- [Background] Cidem M, Karacan I, Diracoglu D, Yildiz A, Kucuk SH, Uludag M, Gun K, Ozkaya M, Karamehmetoglu SS. A Randomized Trial on the Effect of Bone Tissue on Vibration-induced Muscle Strength Gain and Vibration-induced Reflex Muscle Activity. Balkan Med J. 2014 Mar;31(1):11-22. doi: 10.5152/balkanmedj.2013.9482. Epub 2014 Mar 1. PMID 25207162
- [Background] Sebik O, Karacan I, Cidem M, Turker KS. Rectification of SEMG as a tool to demonstrate synchronous motor unit activity during vibration. J Electromyogr Kinesiol. 2013 Apr;23(2):275-84. doi: 10.1016/j.jelekin.2012.09.009. Epub 2012 Oct 23. PMID 23098913